CLINICAL TRIAL: NCT02292173
Title: A Phase 1a/1b Trial of Trametinib in Combination With Sorafenib in Patients With Advanced Hepatocellular Cancer
Brief Title: Trametinib in Combination With Sorafenib in Patients With Advanced Hepatocellular Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17932
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-01

CONDITIONS: Hepatocellular Cancer; Liver Cancer
Keywords: Liver Neoplasms; Liver Diseases; Digestive System Diseases; Advanced; Mitogen-Activated Protein Kinase (MEK) Inhibitor; Kinase Inhibitor
MeSH Terms: conditions — Liver Neoplasms; Liver Diseases; Digestive System Diseases | interventions — trametinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trametinib plus Sorafenib (Experimental): Dose Escalation Followed by Dose Expansion.
  Trametinib: Daily (To start on day 8 during cycle 1 and on day 1 from cycle 2 onwards), according to dose level upon entry.
  Sorafenib: Twice daily, according to dose level upon entry.
  Each cycle is repeated every 28 days.
  Interventions: Drug: Trametinib; Drug: Sorafenib

INTERVENTIONS:
Drug: Trametinib — Dose Escalation:
  Level 1: 1 mg daily. Level 2: 1.5 mg daily. Level 3: 1.5 mg daily. Level 4: 2 mg daily.
  Dose Expansion:
  Maximum Tolerated Dose (MTD)
  Other Names: MEKINIST®
Drug: Sorafenib — Dose Escalation:
  Level 1: 200 mg twice daily. Level 2: 200 mg twice daily. Level 3: 400 mg twice daily. Level 4: 400 mg twice daily.
  Dose Expansion:
  Maximum Tolerated Dose (MTD)
  Other Names: Nexavar®

SUMMARY:
The main purpose of this study is to see whether the combination of trametinib and sorafenib can help people with hepatocellular cancer. Researchers also want to find out if the combination of trametinib and sorafenib is safe and tolerable.

DETAILED DESCRIPTION:
Each cycle will last for 4 weeks. Sorafenib and trametinib will be administered orally on continuous basis. During the first cycle sorafenib will be started on day 1 and trametinib on day 8 to improve tolerance. Participants will get restaging scans every 2 cycles. Participants will continue to receive treatment if they have a stable disease or a better response by Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1.

ELIGIBILITY:
Inclusion Criteria:

* Must have radiographic or histological diagnosis of hepatocellular cancer (HCC), with advanced stage disease that is not amenable to curative surgical resection. Potential participants without histologic diagnosis must meet the radiographic criteria for HCC.
* Child Pugh score must be 5 or 6 (Child Pugh Class A)
* Must have measurable disease by RECIST criteria 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Must have normal organ and marrow function
* Female participants of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male participants must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. For both male and female participants, effective methods of contraception must be used throughout the study and for four months following the last dose.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Participants in the dose expansion part must have tumor that is amenable for biopsy.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Have received radiation therapy, major surgery, other locoregional therapy, within 4 weeks prior to the first dose of study drug
* All prior treatment-related toxicities must be ≤ Grade 1.
* Have received sorafenib or other systemic therapies for treatment of HCC in the past
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception), psychiatric disorder, or other conditions that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures
* History or evidence of cardiovascular risk
* Known history of human immunodeficiency virus (HIV) positivity
* History of retinal vein occlusion (RVO)
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression
* History of interstitial lung disease or pneumonitis
* Are pregnant or lactating
* Any underlying condition that would significantly interfere with the absorption of an oral medication
* History of another active malignancy in last 3 years. Exception: Potential participants who have been disease-free for 3 years, or have a history of completely resected nonmelanoma skin cancer and/or potential participants with indolent second malignancies are eligible.
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; patients with controlled infection or on prophylactic antibiotics are permitted in the study
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide
* Concurrent therapy with approved or investigational anticancer therapy
* Concomitant use of strong Cytochrome P450 3A4 (CYP3A4) inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 18 months
  The MTD for study is defined as the highest dose level at which 1 or less of 6 patients experience a dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria. Further, modified RECIST criteria for HCC will be used to evaluate response. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Response Rate | Up to 3 years
  Response will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria. Further, modified RECIST criteria for HCC will be used to evaluate response. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Overall Survival (OS) | Up to 3 years
  Overall Survival is defined as the time period from start of treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Kim R, Tan E, Wang E, Mahipal A, Chen DT, Cao B, Masawi F, Machado C, Yu J, Kim DW. A Phase I Trial of Trametinib in Combination with Sorafenib in Patients with Advanced Hepatocellular Cancer. Oncologist. 2020 Dec;25(12):e1893-e1899. doi: 10.1634/theoncologist.2020-0759. Epub 2020 Sep 14. PMID 32776632